CLINICAL TRIAL: NCT05581472
Title: Examining Different Components of Online Acceptance and Commitment Therapy for Chronic Pain in a Sample of People With Chiari Malformation
Brief Title: Examining Different Components of Online Acceptance and Commitment Therapy for People With Chiari Malformation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kent State University (Other)
Collaborators: Utah State University (Other); The University of Akron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 270
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain; Chiari Malformation
Keywords: chronic pain; acceptance and commitment therapy; sleep dysfunction; online intervention
MeSH Terms: conditions — Chronic Pain; Arnold-Chiari Malformation; Parasomnias

STUDY DESIGN:
Intervention Model Description: Three groups are created through randomization to either intervention alone, intervention plus phone coaching or the control group. The intervention includes 8 online intervention modules that are administered weekly for 8 weeks. A 7-day sleep diary is administered one week prior to the intervention and one week after the intervention. The control group completes the online sleep diaries and all the same assessments as the treatment group. At the end of the 1 month follow-up they are given the opportunity to receive the intervention.
Who Masked: Outcomes Assessor
Masking Description: Single Blind. Outcome assessor online surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Acceptance and Commitment Therapy Intervention + Phone Coaching (Active Comparator): This online Acceptance and Commitment Therapy intervention is delivered over 8 weeks, in 8 15-minute modules. Additionally, each participant will receive a weekly call for the duration of the intervention (i.e., 9 phone calls: one introduction phone call, 8 module related phone calls) from a Master's-level clinical student who will serve as the participants "phone coach." The intervention includes 8 modules: Away Moves, Letting Go of Control, Noticing Hooks, Stepping Back, Your Values, How You Want to Act, Goal Setting, and Making Commitments). Each module ends with a practice assignment which participants are asked to engage in over the next week.
  During the phone coaching calls, the clinical student will be able to help troubleshoot any technical difficulties being experienced, as well as clarify any questions about the material being taught in the intervention.
  Interventions: Behavioral: Online Acceptance and Commitment Therapy Intervention + Phone Coaching
- Online Acceptance and Commitment Therapy Intervention without phone coaching (Active Comparator): This online Acceptance and Commitment Therapy intervention is delivered over 8 weeks, in 8 15-minute modules. Additionally, each participant will receive a weekly call for the duration of the intervention (i.e., 9 phone calls: one introduction phone call, 8 module related phone calls) from a Master's-level clinical student who will serve as the participants "phone coach." The intervention includes 8 modules: Away Moves, Letting Go of Control, Noticing Hooks, Stepping Back, Your Values, How You Want to Act, Goal Setting, and Making Commitments). Each module ends with a practice assignment which participants are asked to engage in over the next week.
  Interventions: Behavioral: Online Acceptance and Commitment Therapy Intervention without phone coaching
- Waitlist Control (No Intervention): Participants in this arm of the study will complete the same sleep diaries and questionnaires at the same time points as the intervention group, but will not be administered the intervention modules and will not receive any phone coaching. When they have completed the 1-month follow-up they will be offered the intervention.

INTERVENTIONS:
Behavioral: Online Acceptance and Commitment Therapy Intervention + Phone Coaching — The intervention has 8 modules. The modules "Away Moves" and "Letting Go of Control," help to establish creative hopelessness, where one abandons futile struggles against negative internal experiences and accepts new solutions. These two modules also help identify experiential avoidance and focus on acceptance. The modules "Noticing Hooks" and "Stepping Back" focus on diffusion, self as context, and mindfulness. While mindfulness is overtly addressed in the module "Stepping Back", it is weaved through each module. The modules "Your Values" and "How You Want to Act" focus on helping participants identify their values. The modules "Goal Setting" and "Making Commitments" focus on committed action. Each module has a practice assignment which participants are asked to engage in over the next week.
  During the phone coaching calls, the participant will be able to troubleshoot any technical difficulties and ask any questions about the material being taught in the intervention.
  Arms: Online Acceptance and Commitment Therapy Intervention + Phone Coaching
Behavioral: Online Acceptance and Commitment Therapy Intervention without phone coaching — The intervention has 8 modules. The modules "Away Moves" and "Letting Go of Control," help to establish creative hopelessness, where one abandons futile struggles against negative internal experiences and accepts new solutions. These two modules also help identify experiential avoidance and focus on acceptance. The modules "Noticing Hooks" and "Stepping Back" focus on diffusion, self as context, and mindfulness. While mindfulness is overtly addressed in the module "Stepping Back", it is weaved through each module. The modules "Your Values" and "How You Want to Act" focus on helping participants identify their values. The modules "Goal Setting" and "Making Commitments" focus on committed action. Each module has a practice assignment which participants are asked to engage in over the next week.
  Arms: Online Acceptance and Commitment Therapy Intervention without phone coaching

SUMMARY:
Chiari Malformation (CM) is a chronic health condition characterized by brain and spinal malformations and displacements that cause obstruction of cerebrospinal fluid (CSF; Hadley, 2002) circulation. The most common type of CM, CM1, is characterized by the displacement of the cerebellar tonsils more than five millimeters into the foramen magnum (Hadley, 2002). Approximately 215,000 Americans may have CM1, over six times the prevalence of multiple sclerosis (Dilokthornsakul et al., 2016; Speer et al., 2003). Chronic pain is a major problem for patients with CM; (Curone et al., 2017; Garcia et al., 2019). Craniovertebral decompression is the most common surgical intervention for CM1, but it may not be effective in relieving long-term pain and is not recommended for all CM1 patients (Arnautovic et al., 2015; Imperato et al., 2011). In addition to chronic pain, patients with CM also have high levels of depression, anxiety, and sleep dysfunction (Garcia et al., 2019; Lázaro et al., 2018; Watson et al., 2010). Psychological interventions, specifically Acceptance and Commitment Therapy (ACT), have been effective at treating chronic pain when administered online (van de Graaf et al., 2021). We previously found an online self-administered version of ACT to be effective at improving psychological flexibility and chronic pain acceptance in participants with CM (Garcia et al., 2021). In our pilot study (Garcia et al., 2021), participants in the intervention group received phone coaching to improve intervention adherence and use of skills; however, we found that duration of phone coaching did not impact treatment outcomes. We also had excellent retention in the control group. It is unclear whether phone coaching is necessary for treatment engagement or efficacy in groups particularly motivated to seek treatment. If it is not necessary, online ACT can be offered more efficiently and cost-effectively. The proposed study will randomize participants to either ACT+ phone coaching, ACT without coaching, or wait-list control conditions to determine if coaching impacts treatment adherence and outcomes in this population.

Based on power analyses, the sample size will be 111. The sample will be recruited online and randomized to one of the three treatment groups. The intervention will consist of eight modules that are administered weekly over 8 weeks. Follow up assessments will be administered after completion of the intervention, and at one and three months after completion.

DETAILED DESCRIPTION:
Chronic pain is a major problem for patients with CM; over 80% report struggling with neck pain, and 41% report long lasting headaches (Curone et al., 2017; Garcia et al., 2019). Acceptance and Commitment Therapy (ACT) has been widely studied in chronic pain populations using both online and face-to-face modalities (van de Graaf et al., 2021; Veehof et al., 2016). The online intervention for our proposed study was developed by a licensed clinical psychologist and has been tested in a variety of populations (Levin et al., 2020, 2020; Levin, Petersen, et al., 2021). Our prior study found that this intervention was effective at improving psychological flexibility and chronic pain acceptance in participants with CM, the primary mechanisms of ACT (Garcia et al., 2021; Hayes et al., 2006) Moreover, our pilot study indicated that participants were satisfied with the program and found the intervention easy to use with no adverse effects (Garcia et al., 2021). In our prior study, participants in the intervention group received phone coaching designed to improve intervention adherence and use of concepts and skills. This was included based on literature showing a positive impact of coaching on adherence and treatment outcomes in online interventions for mental health outcomes (Mohr et al., 2013; Musiat et al., 2021). Additionally, a recent systematic review of online teletherapy for chronic pain found that interventions with higher levels of therapist guidance were more beneficial and had better adherence (Mariano et al., 2021). However, in our study, we found that duration of phone coaching did not impact treatment outcomes, and another recent study using the same online ACT intervention as our pilot study found no effect of coaching on treatment outcomes, program engagement, or program satisfaction among distressed college students (Levin, Krafft, et al., 2021). Our pilot study also had excellent retention in the wait list control group (85.7%), suggesting that this population is highly motivated to remain engaged. It is unclear whether phone coaching is necessary for treatment engagement, satisfaction, or efficacy in groups particularly motivated to seek treatment. If it is not necessary, online ACT can be offered more efficiently and cost-effectively. The proposed study will randomize participants to either phone coaching or no phone coaching conditions in order to determine the extent to which coaching impacts treatment adherence and outcomes in this population. There will be separate randomization by sex.

The scientific aims are as follows:

Aim One:

Investigate the extent to which phone coaching improves the efficacy of an online ACT intervention for chronic pain.

Hypothesis

1. Participants receiving ACT+ Coaching and ACT only will have increased pain acceptance and psychological flexibility as well as improvement on pain intensity, pain interference, depression, and anxiety than participants in the waitlist control group. We do not expect significant differences between the two treatment groups.

Aim Two:

Identify the effect that ACT has on sleep dysfunction and dysfunctional beliefs and attitudes about sleep.

Hypotheses:

1. Participants receiving ACT+ Coaching and ACT only will have more improvement on dysfunctional beliefs and attitudes about sleep and sleep dysfunction than participants in the waitlist control group. Again, we do not expect significant differences between the two treatment groups.
2. Reduction in sleep dysfunction will be moderated by sleep hygiene practices such that participants with better sleep hygiene will improve in sleep functioning while those with poor sleep hygiene will remain stable or have worsening sleep dysfunction.

The following is a summary of the protocol:

Once recruited, participants will be randomized into the ACT+ coaching group, ACT only group, or the wait-list control. Randomization will be made using an online random number generator. The waitlist control group will receive the same compensation as the intervention groups while in the waitlist control condition. Upon completion of the 8-weeks of questionnaires followed by the 1-month follow up, the waitlist control group will be offered the treatment. Compensation will be in the form of e-gift cards sent to the participant's email, allowing for timely compensation. Compensation will be sent within one week of participants completing each time point.

(Part 1): (Both Treatment & Waitlist Control Groups) Once the participant has signed and submitted the online consent form, they will be asked to complete a set of questionnaires assessing demographics, quality of life, pain interference, pain acceptance, anxiety, depression, stress, and sleep. The survey will take approximately 45 - 60 minutes. Internet access is required to complete these questionnaires on a computer, tablet, or mobile phone.

(Part 2): (Both Treatment & Waitlist Control Groups) Next, participants will be asked to complete a sleep diary daily for 7 days. A Qualtrics link will be emailed to participants each morning (the email will be sent out by midnight the night prior). By clicking on the link, participants will be taken directly to the 2-5-minute survey. Participants are asked to complete this short survey (11 questions) as close to waking as possible to provide the most accurate information. If the participant has not completed the daily diary by noon an additional reminder email will be send out. Once the final day of the sleep diary is completed, participants will be randomly assigned to either the treatment or waitlist control group and will begin on the following Friday. There will be separate randomization by biological sex.

After random assignment, participants will be sent an additional document to sign which contains the specific information about the time commitment for their assigned group. For instance, individuals in the ACT+ coaching group will be informed of the weekly phone call commitment while participants in the ACT only group will not. A participants' signature will be needed in order to proceed with the study.

(Part 3): (Both Treatment Groups) Once a week, for the next 8 weeks, participants will be asked to complete a short battery of questionnaires, followed by the online intervention taking a combined total of approximately 30 - 35 minutes a week. The Qualtrics link will be sent to each participant's email address every Friday morning with the expectation that they will complete the survey and intervention as soon as possible over the next 3 days. If the assessment and intervention has not been completed by the end of day 4 (Monday), participants will receive a phone call to serve as a reminder and to answer any technical or unresolved issues. Each online intervention ends with a practice assignment for the remainder of the week.

(Treatment Group + Phone Coaching) If a participant is assigned to the treatment group with phone coaching, they will receive an email to schedule a 10-15-minute phone call with their "phone coach." The primary goal of the phone coach is to increase adherence to the self-help website (completing web-based sessions and practicing exercises therein). A secondary goal is to support acquisitioning, strengthening and generalization of concepts, exercises and skills taught in the website. However, the role of the phone coach is as a support, not a therapist. The first call will take 10-15 minutes. The goal of this brief "get to know you" phone session is to increase motivation for participating in the self-help program. By the end of the session we'd like to have participants express DARN-C (desire and reasons for, and ability and need to make changes). During this initial phone call the participant will be asked to specify times and days that they are generally available to take the follow-up coaching calls. Follow-up coaching phone calls will take place weekly (8 additional phone calls over the duration of the study) and will last 5-10 minutes. The purpose of the follow up phone calls is to keep participants motivated to use the program and to help them troubleshoot any problems that may interfere with usage. This is also an opportunity to help the participant clarify what about the program is working well for them as well as address any problems. Each participant will then receive a weekly call from a Master's level clinical student; the time of this call will be set up online during the first session in Part 3. During the call the clinical student will be able to help troubleshoot any technical difficulties being experienced, as well as clarify any questions about the material being taught in the intervention.

(Treatment Group without Phone Coaching) If a participant is assigned to the treatment group without phone coaching, they will receive a comprehensive email with instructions for completing the intervention components and weekly surveys. Participants will receive weekly follow up emails and reminders as needed.

(Waitlist Control Group) Each week, for the next 8 weeks, participants will be asked to complete a short battery of questionnaires taking approximately 15 minutes. If any technical difficulties are experienced participants are encouraged to immediately contact chiaristudy@gmail.edu.

(Part 4): (Both Treatment & Waitlist Control Groups) At the beginning of the 9th week, participants will be asked to complete a similar set of questionnaires as in Part 1 excluding the demographic questions. Since the demographic questions will not be asked again, the battery will take approximately 35-40 minutes.

(Part 5): (Both Treatment & Waitlist Control Groups) Next, participants will again be asked to complete a 7- day sleep diary. A Qualtrics link will be emailed to participants each morning (the email will be sent out by midnight the night prior). By clicking on the link, the participants will be taken directly to the 2-5-minute survey. Participants are asked to complete this short survey (11 questions) as close to waking as possible to provide the most accurate information.

(Part 6) (Both Treatment & Waitlist Control Groups) 1-month after completing the intervention participants will be emailed a Qualtrics link to complete the same battery as in Part 4 taking about 35 - 40 minutes.

(Waitlist control group) Upon completion of the 1-month assessment, participants in the waitlist control group will be offered the opportunity to take part in the online intervention.

(Part 7) (Treatment Group only) 3-months after completing the intervention participants will be emailed a Qualtrics link to complete the same battery as in Part 4 and 6 taking about 35 - 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be at least 18 years old, have been diagnosed by a doctor with Chiari Malformation, and report a pain intensity of at least a 3 on a scale from 1-10. If they are taking psychotropic medication participants must be stable on their medication for the past 3 months, and they must have access to the internet. Participants must also be willing to commit approximately an hour a week for 8 weeks to engage in the intervention and homework.

Exclusion Criteria:

Participants will be excluded if they do not speak English, have a sensory impairment (blindness), are less than 18 years old, are without Internet, are not diagnosed with Chiari Malformation, have not experienced persistent pain over the past 3 months, rate their average pain as at least a 3 on a scale from 1-10, have not been stable on psychotropic medication for the past 3 months, are currently receiving therapy or counseling, have active suicidal ideations, and/or have severe psychiatric disorders including bipolar disorder and schizophrenia. Those unstable on medication, having active suicidal ideations, and severe psychiatric disorders will be excluded because they need a higher level of care than will be provided in an online intervention. We are also excluding those currently in therapy because we would not be able to differentiate the impact of the online intervention vs. the impact of their alternative treatment. Participants in the prior ACT pilot study will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in psychological flexibility over time measured by the Acceptance and Action Questionnaire (AAQ). | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.
  The seven AAQ Items are scored on a scale from 1 (never true) to 7 (always true). Lower scores on this scale indicate greater psychological flexibility, the core mechanism of Acceptance and Commitment Therapy (Bond et al., 2011; Hayes et al., 2006).
Change in chronic pain acceptance over time assessed by the Chronic Pain Acceptance Questionnaire-Revised (CPAQ). | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.
  The CPAQ is a 20-item scale that assesses acceptance of chronic pain-related thoughts, feelings, and experiences (McCracken et al., 2004). Questions are on a Likert scale ranging from 0 (never true) to 6 (always true). While the total score is indicative of broader acceptance of chronic pain, two subscales have been empirically identified to predict pain-related disability and distress: activities engagement and pain willingness (McCracken et al., 2004; Vowles et al., 2008).
Change in pain intensity over time as assessed with the Numeric Rating Scale (NRS). | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.]
  The NRS has individuals rate their pain from 0 (no pain) to 10 (worst pain imaginable) on four separate time anchors: pain right now, usual level of pain during the last week, best level of pain during the last week, and worst level of pain during the last week (Jensen et al., 1999). Due to a lack of clear consensus on which time anchor to use, all 4 items will be examined separately (Patel et al., 2021).
Change in pain interference over time assessed by the pain interference subscale of the Brief Pain Inventory. | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.
  The 7-item pain interference subscale asks participants to rate how much pain has interfered with their general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life (Cleeland, 2009). Ratings are on a scale of 0 ("Does not interfere") to 10 ("Completely Interferes").
Change in symptoms of depression and anxiety over time assessed by the Depression, Anxiety, and Stress Scale (DASS-21). | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.
  The Depression, Anxiety and Stress Scale (DASS-21) is a 21-item scale that assesses depression, anxiety, and stress (Lovibond & Lovibond, 1995). The 21 items of the DASS-21 are rated on a scale of 0 ("Did not apply to me at all") to 3 ("Applied to me very much of the time.")

SECONDARY OUTCOMES:
Change in sleep dysfunction assessed by the Sleep Diary. | Assessed at baseline and at the 1 week follow up after the intervention.
  The 7-day sleep diary is a 14-item measure comprised of the 8-question Consensus Sleep Diary core which assesses sleep onset latency, quantity, and quality of sleep; we also added one item to ask participants to estimate how long they slept (Carney et al., 2012). The sleep diary also included 4 additional questions asking participants to rate their arousal, nervousness, feelings of restlessness, pain and mood on a scale of 0 ("Not at all) to 10 ("a lot;" Tang et al., 2012).
Change in sleep dysfunction over time assessed by the Insomnia Severity Index. | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.
  The Insomnia Severity Index is a 7-item questionnaire that assesses sleep quality and dysfunction. Items are rated on a scale of 0 ("None" or "Not at all interfering") to 4 ("Very Severe" or "Very much interfering;" (Morin et al., 2011)
Change in dysfunctional beliefs and attitudes about sleep over time assessed by the Dysfunctional Beliefs and Attitudes about Sleep questionnaire (DBAS)-16. | Assessed at baseline, 8 intervention weeks, 1 week follow up, 1 month follow up, and three month follow up.]
  The DBAS is a 16-item questionnaire that assesses the extent to which participants agree with negative or dysfunctional beliefs about sleep. The items are rated on a scale of 0 ("Strongly Disagree") to 10 (Strongly agree") and the items are designed to capture the cognitive component of insomnia (Morin et al., 2007).
Percentage of participants who met criteria for Minimal Clinically Important Difference (MCID) in pain scores. | MCID will be calculated for baseline-1 week post intervention, baseline-1 month post intervention, and baseline-3 months post intervention.]
  A minimum of 20% decrease in pain ratings (2-point reduction) will indicate minimum change while a substantial pain reduction will be defined as a 50% or greater decrease (5-point reduction). Pain intensity MCID will be calculated on the 4 NRS pain intensity items individually. For pain interference, a minimum of 1 point decrease will be needed on the pain interference subscale of the Brief Pain inventory (Dworkin et al., 2008; Smith et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Delahanty, PhD, Principal Investigator — Kent State University
Locations (1):
- Kent state University, Kent, Ohio, United States

REFERENCES:
- [Background] Arnautovic A, Splavski B, Boop FA, Arnautovic KI. Pediatric and adult Chiari malformation Type I surgical series 1965-2013: a review of demographics, operative treatment, and outcomes. J Neurosurg Pediatr. 2015 Feb;15(2):161-77. doi: 10.3171/2014.10.PEDS14295. Epub 2014 Dec 5. PMID 25479580
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Curone M, Valentini LG, Vetrano I, Beretta E, Furlanetto M, Chiapparini L, Erbetta A, Bussone G. Chiari malformation type 1-related headache: the importance of a multidisciplinary study. Neurol Sci. 2017 May;38(Suppl 1):91-93. doi: 10.1007/s10072-017-2915-8. PMID 28527081
- [Background] Dilokthornsakul P, Valuck RJ, Nair KV, Corboy JR, Allen RR, Campbell JD. Multiple sclerosis prevalence in the United States commercially insured population. Neurology. 2016 Mar 15;86(11):1014-21. doi: 10.1212/WNL.0000000000002469. Epub 2016 Feb 17. PMID 26888980
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Garcia MA, Allen PA, Li X, Houston JR, Loth F, Labuda R, Delahanty DL. An examination of pain, disability, and the psychological correlates of Chiari Malformation pre- and post-surgical correction. Disabil Health J. 2019 Oct;12(4):649-656. doi: 10.1016/j.dhjo.2019.05.004. Epub 2019 May 21. PMID 31147250
- [Background] Hadley DM. The Chiari malformations. J Neurol Neurosurg Psychiatry. 2002 Jun;72 Suppl 2(Suppl 2):ii38-ii40. doi: 10.1136/jnnp.72.suppl_2.ii38. No abstract available. PMID 12122202
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Imperato A, Seneca V, Cioffi V, Colella G, Gangemi M. Treatment of Chiari malformation: who, when and how. Neurol Sci. 2011 Dec;32 Suppl 3:S335-9. doi: 10.1007/s10072-011-0709-y. PMID 21822700
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Levin ME, Krafft J, Davis CH, Twohig MP. Evaluating the effects of guided coaching calls on engagement and outcomes for online acceptance and commitment therapy. Cogn Behav Ther. 2021 Sep;50(5):395-408. doi: 10.1080/16506073.2020.1846609. Epub 2021 Jan 12. PMID 33433264
- [Background] Levin ME, Krafft J, Hicks ET, Pierce B, Twohig MP. A randomized dismantling trial of the open and engaged components of acceptance and commitment therapy in an online intervention for distressed college students. Behav Res Ther. 2020 Mar;126:103557. doi: 10.1016/j.brat.2020.103557. Epub 2020 Jan 22. PMID 32014692
- [Background] Levin ME, Petersen JM, Durward C, Bingeman B, Davis E, Nelson C, Cromwell S. A randomized controlled trial of online acceptance and commitment therapy to improve diet and physical activity among adults who are overweight/obese. Transl Behav Med. 2021 Jun 17;11(6):1216-1225. doi: 10.1093/tbm/ibaa123. PMID 33289785
- [Background] Mariano TY, Wan L, Edwards RR, Jamison RN. Online teletherapy for chronic pain: A systematic review. J Telemed Telecare. 2021 May;27(4):195-208. doi: 10.1177/1357633X19871746. Epub 2019 Sep 5. PMID 31488004
- [Background] McCracken LM, Vowles KE, Eccleston C. Acceptance of chronic pain: component analysis and a revised assessment method. Pain. 2004 Jan;107(1-2):159-66. doi: 10.1016/j.pain.2003.10.012. PMID 14715402
- [Background] Mohr DC, Duffecy J, Ho J, Kwasny M, Cai X, Burns MN, Begale M. A randomized controlled trial evaluating a manualized TeleCoaching protocol for improving adherence to a web-based intervention for the treatment of depression. PLoS One. 2013 Aug 21;8(8):e70086. doi: 10.1371/journal.pone.0070086. eCollection 2013. PMID 23990896
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Morin CM, Vallieres A, Ivers H. Dysfunctional beliefs and attitudes about sleep (DBAS): validation of a brief version (DBAS-16). Sleep. 2007 Nov;30(11):1547-54. doi: 10.1093/sleep/30.11.1547. PMID 18041487
- [Background] Musiat P, Johnson C, Atkinson M, Wilksch S, Wade T. Impact of guidance on intervention adherence in computerised interventions for mental health problems: a meta-analysis. Psychol Med. 2022 Jan;52(2):229-240. doi: 10.1017/S0033291721004621. Epub 2021 Nov 22. PMID 34802474
- [Background] Patel KV, Amtmann D, Jensen MP, Smith SM, Veasley C, Turk DC. Clinical outcome assessment in clinical trials of chronic pain treatments. Pain Rep. 2021 Jan 21;6(1):e784. doi: 10.1097/PR9.0000000000000784. eCollection 2021 Jan-Feb. PMID 33521482
- [Background] Smith SM, Dworkin RH, Turk DC, McDermott MP, Eccleston C, Farrar JT, Rowbotham MC, Bhagwagar Z, Burke LB, Cowan P, Ellenberg SS, Evans SR, Freeman RL, Garrison LP, Iyengar S, Jadad A, Jensen MP, Junor R, Kamp C, Katz NP, Kesslak JP, Kopecky EA, Lissin D, Markman JD, Mease PJ, O'Connor AB, Patel KV, Raja SN, Sampaio C, Schoenfeld D, Singh J, Steigerwald I, Strand V, Tive LA, Tobias J, Wasan AD, Wilson HD. Interpretation of chronic pain clinical trial outcomes: IMMPACT recommended considerations. Pain. 2020 Nov;161(11):2446-2461. doi: 10.1097/j.pain.0000000000001952. PMID 32520773
- [Background] Speer MC, Enterline DS, Mehltretter L, Hammock P, Joseph J, Dickerson M, Ellenbogen RG, Milhorat TH, Hauser MA, George TM. Review Article: Chiari Type I Malformation with or Without Syringomyelia: Prevalence and Genetics. J Genet Couns. 2003 Aug;12(4):297-311. doi: 10.1023/A:1023948921381. PMID 26141174
- [Background] Tang NK, Goodchild CE, Sanborn AN, Howard J, Salkovskis PM. Deciphering the temporal link between pain and sleep in a heterogeneous chronic pain patient sample: a multilevel daily process study. Sleep. 2012 May 1;35(5):675-87A. doi: 10.5665/sleep.1830. PMID 22547894
- [Background] van de Graaf DL, Trompetter HR, Smeets T, Mols F. Online Acceptance and Commitment Therapy (ACT) interventions for chronic pain: A systematic literature review. Internet Interv. 2021 Oct 1;26:100465. doi: 10.1016/j.invent.2021.100465. eCollection 2021 Dec. PMID 34660209
- [Background] Veehof MM, Trompetter HR, Bohlmeijer ET, Schreurs KM. Acceptance- and mindfulness-based interventions for the treatment of chronic pain: a meta-analytic review. Cogn Behav Ther. 2016;45(1):5-31. doi: 10.1080/16506073.2015.1098724. Epub 2016 Jan 28. PMID 26818413
- [Background] Vowles KE, McCracken LM, McLeod C, Eccleston C. The Chronic Pain Acceptance Questionnaire: confirmatory factor analysis and identification of patient subgroups. Pain. 2008 Nov 30;140(2):284-291. doi: 10.1016/j.pain.2008.08.012. Epub 2008 Sep 27. PMID 18824301
- [Derived] Rabinowitz EP, Ripley GH, Lemek C, Allen PA, Delahanty DL. High levels of patient self advocacy may confound clinical research in understudied patient populations. J Health Psychol. 2025 Sep;30(10):2816-2822. doi: 10.1177/13591053241286643. Epub 2024 Sep 30. PMID 39345001
- See also: Lázaro, 2018 — https://doi.org/10.31083/j.jin.2018.04.0414
- See also: Lovibond 1995 — https://books.google.com/books/about/Manual_for_the_Depression_Anxiety_Stress.html?id=mXoQHAAACAAJ
- See also: Watson, 2010 — https://link.springer.com/article/10.1111/j.1479-8425.2010.00456.x